CLINICAL TRIAL: NCT06282094
Title: ViSiGi LUX Bariatric Sizing and Calibration System Usability Study
Brief Title: ViSiGi LUX Bariatric Sizing and Calibration System
Status: Recruiting | Type: Observational
Sponsor: Boehringer Labs LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: LUX
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the new ViSiGi LUX.

DETAILED DESCRIPTION:
ViSiGi is used during numerous gastric and bariatric procedures. The new device, ViSiGi LUX functions as the FDA-cleared ViSiGi but has the added visualization of NIR lights.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able to consent
* candidate for robotic bariatric surgery

Exclusion Criteria:

* esophageal stricture that does not allow passage of the device
* conditions that would preclude gastric or bariatric surgical procedures
* pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing gastric or bariatric procedures.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Physician Feedback | 6 months
  The physician provides feedback and comments on the usability of the device. The physician will rate the device on a Likert scale. 1-7 higher score is better

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No